CLINICAL TRIAL: NCT03919773
Title: IVIG (Gamunex-C) Study of Treatment for Autoimmune Neuropathic Dysautonomia/Postural Tachycardia (POTS)
Brief Title: IVIG (Gamunex-C) Treatment Study for POTS Subjects
Acronym: iSTAND
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Grifols Biologicals, LLC (Industry); Dysautonomia International (Other)
Responsible Party: Principal Investigator, Steven Vernino MD PhD, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2018-0005
Record Dates: First submitted 2019-02-05; First posted 2019-04-18 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Postural Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Immunoglobulins, Intravenous; Albumins

STUDY DESIGN:
Intervention Model Description: double-blind randomized controlled crossover pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment IVIG Arm (Active Comparator): IVIG (Gammunex-C) infusion (0.4 gm/kg) every week for 4 weeks, then every 2 weeks for 8 weeks (12 weeks total).
  Interventions: Drug: IVIG
- Treatment Albumin Arm (Placebo Comparator): albumin infusion (0.4 gm/kg) every week for 4 weeks then every 2 weeks for 8 weeks (12 weeks total) during
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: IVIG — If you participate in this study there will be 18 scheduled treatment infusions during the 30 week study period. All the study visits and treatment visits will be outpatient visits.
  Once you qualify to participate in the study and begin treatment, there will be two 12 week treatment periods separated by a 6 week washout period. The infusion visits will take approximately 3-4 hours each.
  Other Names: intravenous immunoglobulin
  Arms: Treatment IVIG Arm
Drug: Albumin — This will be the matching placebo used in the study.
  Arms: Treatment Albumin Arm

SUMMARY:
The purpose of this trial is to evaluate the symptomatic benefits of immunomodulatory treatment with IVIG for POTS (postural tachycardia syndrome) patients with evidence of autoimmunity.

DETAILED DESCRIPTION:
Gammunex-C, a form of intravenous immunoglobulin (IVIG), is approved for the treatment of chronic inflammatory demyelinating neuropathy (CIDP) or idiopathic thrombocytopenic purpura (ITP). IVIG has been in use for many decades in the treatment of these disorders and many other inflammatory/autoimmune diseases. It is generally very safe and well tolerated. More recently, IVIG has been proposed as an effective treatment for presumed inflammatory neurological disorders which do not meet the criteria for CIDP. Specifically, case reports and cases series have indicated therapeutic responses to IVIG in autonomic neuropathies.

Intravenous Albumin is approved for the treatment of hypovolemia (see attached package insert). The use of albumin to increase plasma volume in patients with POTS has been suggested. In this study, albumin will be used as an active control treatment to provide the same volume and protein load as IVIG but without the immunomodulatory effects.

There have been few well designed clinical therapy trials aimed at POTS patients and even fewer that are aimed at a particular pathophysiological subtype of POTS. Evidence suggests that POTS is a heterogeneous disorder with differing underlying mechanisms. Several uncontrolled case series have suggested a benefit of IVIG for POTS, but the volume expansion associated with infusion of IVIG make it difficult to assess the immunomodulatory effects of this treatment. We propose to evaluate the efficacy of IVIG using a double-blind randomized cross over design that will determine efficacy while reducing effects of inter-subject variability and placebo effect which are common problems in POTS therapy research. Even with the statistical advantages of a crossover design, the treatment cohort will be small, and this study is designed to be a pilot (phase II) study to evaluate the feasibility, tolerability and potential benefits of treatment. The results of this pilot study will provide the impetus and rationale for a larger multicenter clinical trial to definitively evaluate immunomodulatory treatment in POTS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, and able to provide informed consent
* Diagnosis of POTS (see Table 1)
* COMPASS-31 symptom score showing moderate to severe autonomic symptoms
* At least 3 of the following clinical or laboratory features of autoimmunity

  * One or more serum autoantibodies (ANA ≥ 1:160, gAChR antibody > 0.2 nmol/L, positive ENA, aPL, TTG, gliadin) or inflammatory markers (ESR > 30, CRP > 2, low C3 complement or low immunoglobulin IgG level)
  * Confirmed personal history or family history of defined autoimmune disease including Hashimoto's thyroiditis, celiac disease, antiphospholipid syndrome, rheumatoid arthritis, SLE, or Sjogren's syndrome
  * Clear history of acute or subacute onset following infection, immunization, injury/concussion, surgery or pregnancy.
  * Evidence of esophageal, gastric or intestinal dysmotility (with weight loss)
  * Evidence of small fiber neuropathy (abnormal QSART or IENFD)
* Stable oral medical therapy for past 3 months
* Ambulatory at time of screening

Exclusion Criteria:

* Current or previous immunosuppression therapy or IVIG treatment
* Contraindication to intravenous immunoglobulin or intravenous albumin
* Known allergic reactions to blood products including intravenous immunoglobulin (IVIG) and/or subcutaneous immunoglobulin (SCIG), such as history of clinically relevant hemolysis after IVIG infusion, aseptic meningitis, recurrent severe headache, hypersensitivity, severe generalized or severe local skin reaction.
* Inadequate peripheral venous access
* Evidence of renal insufficiency (Cr > 1.5 x elevated) or liver disease (transaminases > 2.5x upper limit) at screening
* History of thrombotic episode within 3 years of enrollment
* Other major medical issue which, in investigators opinion, increases risk for adverse event over the next 12 months or may require separate management.
* Female patients who are premenopausal and are (a) pregnant based on serum pregnancy test, or (b) breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Vernino, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All patient information will be de-identified if sent out. Any AE and/or SAE will be sent out for review.

REFERENCES:
- [Background] Goodman BP, Crepeau A, Dhawan PS, Khoury JA, Harris LA. Spectrum of Autonomic Nervous System Impairment in Sjogren Syndrome. Neurologist. 2017 Jul;22(4):127-130. doi: 10.1097/NRL.0000000000000134. PMID 28644253

RESULTS

PARTICIPANT FLOW:
Groups:
- IVIG First, Then Albumin: Once qualified for the study and starting treatment, there are two 12 week treatment periods separated by a 6 week washout period. The infusion visits will take approximately 3-4 hours each. All the study visits and treatment visits are outpatient visits.
  Treatment period 1: IVIG (Gammunex-C) infusion (0.4 gm/kg) every week for 4 weeks, then every 2 weeks for 8 weeks (12 weeks total, 8 infusions).
  Washout period: 6 weeks
  Treatment period 2: Albumin infusion: (0.4 gm/kg) every week for 4 weeks then every 2 weeks for 8 weeks (12 weeks total, 8 infusions). This will be the matching control treatment used in the study.
- Albumin First, Then IVIG: Once qualified for the study and starting treatment, there are two 12 week treatment periods separated by a 6 week washout period. The infusion visits will take approximately 3-4 hours each. All the study visits and treatment visits are outpatient visits.
  Treatment period 1: Albumin infusion: (0.4 gm/kg) every week for 4 weeks then every 2 weeks for 8 weeks (12 weeks total, 8 infusions). This will be the matching control treatment used in the study.
  Washout period: 6 weeks
  Treatment period 2: IVIG (Gammunex-C) infusion (0.4 gm/kg) every week for 4 weeks, then every 2 weeks for 8 weeks (12 weeks total, 8 infusions).
Period: First Intervention- (12 Weeks)
Arm/Group | IVIG First, Then Albumin | Albumin First, Then IVIG
Started | 16 | 14
Completed | 15 | 12
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 1
Period: Washout (6 Weeks)
Arm/Group | IVIG First, Then Albumin | Albumin First, Then IVIG
Started | 15 | 12
Completed | 12 | 12
Not Completed | 3 | 0
Period: Second Intervention-(12 Weeks)
Arm/Group | IVIG First, Then Albumin | Albumin First, Then IVIG
Started | 12 | 12
Completed | 10 | 11
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVIG First, Then Albumin | Albumin First, Then IVIG | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (8.75) | 31.9 (9.99) | 31.8 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30
Time since symptom onset (years), median (IQR) [Median (Inter-Quartile Range); unit: years] | 4.0 [2.0 to 6.5] | 4.0 [2.0 to 8.0] | 4.0 [2.0 to 7.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptoms Measured by Change in COMPASS-31 Score (After Initial Treatment Phase)
Description: Primary outcome was change in autonomic symptom burden, assessed by total COMPASS-31 (sum of scaled subscores), comparing assessment at week 13 (2 weeks after final infusion) minus the assessment at baseline. This questionnaire generates a weighted score from 0 to 100, and questions fall into one of six domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor function. A COMPASS-31 (Composite Autonomic Symptom Score-31) score of ≥20 suggests moderate-to-severe autonomic dysfunction.
  Higher scores indicate more severe symptoms. A reduction in score (negative change over time) indicates better outcome or response to treatment.
Time Frame: Baseline,13 weeks
Population: The primary outcome measure was assessed only during the first treatment phase and hence, only 15 participants who received IVIG treatment and 13 participants who received Albumin treatment were analyzed for this primary outcome measure. The 1 patient (Albumin- First intervention group) who was a protocol violation was included in the analysis. The 2 patients (1 each from IVIG and Albumin- first intervention groups) with SAEs were not included in the analysis since lost to follow-up.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Treatment IVIG Arm: IVIG (Gammunex-C) infusion (0.4 gm/kg) every week for 4 weeks, then every 2 weeks for 8 weeks (12 weeks total).
  IVIG: If you participate in this study there will be 18 scheduled treatment infusions during the 30 week study period. All the study visits and treatment visits will be outpatient visits.
  Once you qualify to participate in the study and begin treatment, there will be two 12 week treatment periods separated by a 6 week washout period. The infusion visits will take approximately 3-4 hours each.
Arm/Group | Treatment IVIG Arm | Treatment Albumin Arm
Number analyzed (Participants) | 15 | 13
score on a scale | -5.5 [-27 to 21] | -10.6 [-28 to 2]
Statistical Analysis 1: Comparison: Treatment IVIG Arm vs Treatment Albumin Arm; Intention-to-treat analysis; Test type: Superiority; p = 0.629, Kruskal-Wallis

2. Secondary Outcome: Number of Participants With Clinical Improvement
Description: The count of participants with clinical improvement at 13 weeks is being reported here. Clinical improvement was defined as a reduction of the COMPASS-31 total score by 20% or more. Lower scores are associated with improvement and a 20% reduction was used as a meaningful change in previous studies of POTS
Time Frame: 13 weeks
Population: The secondary outcome measure was assessed only for the first treatment phase and hence, only 15 participants who received IVIG treatment and 13 participants who received Albumin treatment were analyzed for this outcome measure. The 1 patient (Albumin- First intervention group) who was a protocol violation was included in this analysis . The 2 patients (1 each from IVIG and Albumin- first intervention groups) with SAEs were not included in the analysis since lost to follow-up.
Measure: Number; unit: participants
Arm/Group | Treatment IVIG Arm | Treatment Albumin Arm
Number analyzed (Participants) | 15 | 13
participants | 7 | 5
Statistical Analysis 1: Comparison: Treatment IVIG Arm vs Treatment Albumin Arm; comparison of proportion with positive treatment response (as defined) in IVIG group compared to albumin; Test type: Superiority; p = 0.718, Fisher Exact

ADVERSE EVENTS:
Time Frame: 30 weeks
Arm/Group | Treatment IVIG Arm | Treatment Albumin Arm
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/28 | 2/26
Other Adverse Events (participants affected / at risk) | 25/28 | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment IVIG Arm (N=28) | Treatment Albumin Arm (N=26)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Pneumonia requiring hospitalization
Magnetic resonance imaging of head abnormal (finding) (Nervous system disorders) | 1 (1) | 0 (0) — Abnormal MRI during evaluation of headache
Severe Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ovarian Cyst rupture (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment IVIG Arm (N=28) | Treatment Albumin Arm (N=26)
Headache (Nervous system disorders) | 18 (18) | 14 (14)
Fatigue (General disorders) | 8 (8) | 9 (9)
Pain (General disorders) | 8 (8) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)
gastrointestinal symptom (Gastrointestinal disorders) | 6 (6) | 5 (5)
Fever (General disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03919773/Prot_001.pdf
  • Statistical Analysis Plan (2023-10-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT03919773/SAP_002.pdf